CLINICAL TRIAL: NCT05933278
Title: Immunogenicity & Safety of IndoVac® as a Homologous Booster Dose Against COVID-19 in Adults Aged 18 Years and Above in Indonesia
Brief Title: Homologous Booster Study of COVID-19 Protein Subunit Recombinant Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PT Bio Farma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CoV2-Booster 0323
Record Dates: First submitted 2023-07-05; First posted 2023-07-06 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: COVID-19
Keywords: COVID-19 vaccine; Booster
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants who previously completed primary doses of vaccine (Experimental): Participants who previously completed primary doses of vaccine
  Interventions: Biological: SARS-CoV-2 Subunit Recombinant Protein Vaccine

INTERVENTIONS:
Biological: SARS-CoV-2 Subunit Recombinant Protein Vaccine — SARS-CoV-2 RBD subunit recombinant protein, manufactured by PT Bio Farma

SUMMARY:
Open-label, prospective intervention study of IndoVac® as a single, homologous booster dose

DETAILED DESCRIPTION:
This trial is open-label, prospective intervention study. A total of 150 subjects who had previously received complete primary doses of IndoVac® in phase III and are willing to participate in the study by signing the consent form, will be involved in this trial. The regimen of the vaccine 0.5 ml injected as a single booster dose.

Evaluation will be conducted for safety and immunogenicity for all subjects. Safety evaluation include AEs until 28 days post booster dose, with AESIs and SAEs throughout the trial. Immunogenicity evaluation will compare pre-booster antibody titer (baseline) to post- booster antibody titer at 14 days, 28 days, 3 months, 6 months, and 12 months timepoint. Interim evaluation will be performed at 14 days post booster dose for Emergency Use Authorization (EUA) consideration. All subjects will be followed up until 12 months post booster dose.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically healthy subjects aged 18 years and above.
2. Subjects had previously received complete primary doses of IndoVac® with the last dose administered minimum 12 months but no longer than 18 months prior to inclusion.
3. Subjects have been informed properly regarding the study and signed the informed consent form.
4. Subjects will commit to comply with the instructions of the investigator and the schedule of the trial.

Exclusion Criteria:

1. Subjects concomitantly enrolled or scheduled to be enrolled in another trial.
2. Subjects had received booster dose of COVID-19 vaccine.
3. History of COVID-19 within 3 months prior to enrollment (based on anamnesis or other examinations).
4. Evolving mild, moderate, or severe illness, especially infectious disease, or fever (body temperature ≥37.5°C, measured with infrared thermometer/thermal gun).
5. Women who are pregnant or planning to become pregnant during the study period (judged by self- report of subjects and urine pregnancy test results).
6. History of uncontrolled asthma, allergy to vaccines or vaccine ingredients, and severe adverse reactions to vaccines, such as urticaria, dyspnea, and angioneurotic edema.
7. History of uncontrolled coagulopathy or blood disorders contraindicating intramuscular injection.
8. Patients with serious chronic diseases (serious cardiovascular diseases, uncontrolled hypertension or diabetes, liver or kidney diseases, malignant tumors, etc.) which according to the investigator might interfere with the assessment of the trial objectives.
9. History of confirmed or suspected immunosuppressive or immunodeficient state or in the previous 4 weeks had received a treatment likely to alter the immune response (intravenous immunoglobulins, blood-derived products, or long- term corticosteroid therapy (> 2 weeks)).
10. History of uncontrolled epilepsy or other progressive neurological disorders, such as Guillain- Barre Syndrome.
11. Subjects had received any vaccination (other than COVID-19 vaccine) within 1 month before IP immunization.
12. Subjects plan to move from the study area before the end of study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2023-07-25 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-09-05 (Actual)

PRIMARY OUTCOMES:
Neutralizing antibody before and at 14 days after booster dose | Baseline, 14 days after booster dose
  Geometric Mean Titer (GMT) and Geometric Mean Fold Ratio (GMFR) of SARS-CoV-2 neutralizing antibody against Omicron variant

SECONDARY OUTCOMES:
Neutralizing antibody at 28 days after booster dose | Baseline, 14 days, 28 days after booster dose
  Geometric Mean Titer (GMT) and Geometric Mean Fold Ratio (GMFR) of SARS-CoV-2 neutralizing antibody against Omicron variant
RBD-binding IgG antibody before, at 14 days and 28 days after booster dose | Baseline, 14 days, 28 days after booster dose
  Geometric Mean Titer (GMT) and Geometric Mean Fold Ratio (GMFR) of SARS-CoV-2 RBD-binding IgG antibody
Antibody persistence at 3, 6, and 12 months after booster dose | Baseline, 3 months, 6 months, 12 months after booster dose
  Geometric Mean Titer (GMT) and Geometric Mean Fold Ratio (GMFR) of SARS-CoV-2 RBD-binding IgG antibody
Safety after booster dose | Baseline to 12 months after booster dose
  Number and percentage of subjects with solicited and unsolicited Adverse Events (AEs), Serious Adverse Events (SAEs), Adverse Events of Special Interest (AESIs)

CONTACTS AND LOCATIONS:
Overall Officials: Yetty Movieta Nency, MD, Principal Investigator — Faculty of Medicine Universitas Diponegoro
Locations (1):
- Faculty of Medicine Diponegoro University, Semarang, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: No